CLINICAL TRIAL: NCT02116569
Title: A Phase I Study of JNJ-54761414 (Daratumumab) in Japanese Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of Daratumumab in Japanese Participants With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR104072; 54767414MMY1002 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Daratumumab; JNJ-54767414; Phase 1; Relapse; Refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daratumumab 8 milligram per kilogram (mg/kg) (Experimental): Participants will be administered intravenously with daratumumab at a dose of 8 mg/kg up to 8 weeks (total 7 infusions). After 8 weeks, participants will receive daratumumab intravenously two times in every 2 weeks until Week 24 followed by one time in 4 weeks until study discontinuation.
  Interventions: Drug: Daratumumab
- Daratumumab 16 mg/kg (Experimental): Participants will be administered intravenously with daratumumab at a dose of 16 mg/kg up to 8 weeks (total 7 infusions). After 8 weeks, participants will receive daratumumab intravenously at a same dose, two times in every 2 weeks until Week 24 followed by one time in 4 weeks until study discontinuation.
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Participants will be administered intravenously with daratumumab at a dose of 8 or 16 mg/kg up to 8 weeks (total 7 infusions). After 8 weeks, participants will receive daratumumab intravenously at a same dose, two times in every 2 weeks until Week 24 followed by one time in 4 weeks until study discontinuation. If the dose exceeds 24 mg/kg, then it will be considered as overdose in this study.
  Other Names: JNJ-54767414

SUMMARY:
The purpose of this study is to evaluate the tolerability and safety of Daratumumab in Japanese participants with relapsed (the return of a medical problem) or refractory (not responding to treatment) multiple myeloma (cancer of plasma cells in bone marrow, characterized by the presence of abnormal proteins in the blood).

DETAILED DESCRIPTION:
This is a Phase 1, open-label (all participants and study personnel will know the identity of the study treatments) and multicenter (study conducted at multiple sites) study in Japanese participants. The study will include a Screening Phase, a Treatment Phase, and a Follow-up Phase. The Treatment Phase consists of 2 parts: intense dosing regimen and less intense dosing regimen. Follow-up phase will be until 8 weeks after last dose administration/death/lost to follow up/consent withdrawal for study participation or study end, whichever occurs first. The primary endpoints will be Dose Limiting Toxicity (DLTs) and overall Adverse Events (AEs) profiling. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants proven to have symptomatic (having symptoms) multiple myeloma according the International Myeloma Working Group (IMWG) diagnostic criteria
* Participant must have measurable disease defined by either or both the following measurements: a) Serum M-protein greater than or equal to (>=) 1 gram per deciliter (g/dL) (>=10 gram per liter [g/L]) (except for serum immunoglobulin A [IgA] M-protein >= 0.5 g/dL); b) Urine M-protein >=200 milligram per 24 hour (mg/24 h); in case immunoglobulin D [IgD] or immunoglobulin E [IgE] M-protein, quantification should be performed
* Participant must have relapsed or refractory multiple myeloma after receiving at least 2 previous therapies, and without further established treatment options
* Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Participant must have life expectancy greater than (>) 3 months

Exclusion Criteria:

* Participant has received daratumumab or other anti-cluster of differentiation 38 (anti-CD38) therapies previously
* Participant has received anti-myeloma treatment within 2 weeks before administration of the study drug
* Participant has previously received an allogenic stem cell transplant; or participant has received autologous stem cell transplantation (ASCT) within 12 weeks before administration of the study drug
* Participant has a history of malignancy (other than multiple myeloma) within 5 years before administration of the study drug
* Participant is exhibiting clinical signs of meningeal involvement of multiple myeloma

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicities (DLT) | Day 1 up to Day 36
  The Dose-Limiting Toxicities (DLTs) are based on drug-related adverse events and defined as any of the following events: Infusion-related reactions, non-hematologic toxicity of Grade 3 or higher, or hematologic toxicity.
Number of Participants affected by Adverse Events | Baseline up to 4 Weeks after the last dose of study drug administration
  An AE is any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

SECONDARY OUTCOMES:
Percentage of Participants With Overall Response | Baseline until disease progression, unmanageable adverse event or death, whichever occurs first, up to 1 year
  The Overall Response rate is defined according to Internal Myeloma Working Group criteria based on participants achieving greater than or equal to (>=) partial Response, including participants achieving stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR). Percentage of participants with overall response will be reported.
Time to Response | Baseline until first documented response or up to 1 year
  Time to response is defined as the time from the date of first dose of study treatment to the date of the first documentation of observed response.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (2):
- Japan (2):
  - Nagoya
  - Tokyo

REFERENCES:
- [Derived] Li X, Dosne AG, Perez Ruixo C, Perez Ruixo JJ. Pharmacodynamic-Mediated Drug Disposition (PDMDD) Model of Daratumumab Monotherapy in Patients with Multiple Myeloma. Clin Pharmacokinet. 2023 May;62(5):761-777. doi: 10.1007/s40262-023-01232-8. Epub 2023 Apr 6. PMID 37022569
- See also: A Phase 1 Study of JNJ-54767414 (Daratumumab) in Japanese Patients With Relapsed or Refractory Multiple Myeloma — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=6838&filename=54767414MMY1002_Synopsis.pdf